CLINICAL TRIAL: NCT00462371
Title: Open-Label, Randomised Trial Comparing Efficacy of Continuous Subcutaneous Insulin Infusion(CSII) and Multiple Daily Insulin Injections (MDII) in Improving Glycemic Control and Quality of Life in Poorly Regulated Type 1 Diabetic Children.
Brief Title: Comparison Between Insulin Pump Treatment and Multiple Daily Insulin Injections in Diabetic Type 1 Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Ministry of Health (Ambiguous)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASB21004821
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus, Type 1; Child
Keywords: quality of life; child diabetes mellitus type 1; Continuous subcutaneous insulin infusion(CSII); metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Insulin pump (CSII)

SUMMARY:
Comparison between insulin pump treatment and multiple daily insulin injections in 38 children with type 1 diabetes4-16 years old. Outcome metabolic control, quality of life, impact of disease and cost effectiveness.

We hypothesised that insulin pump treatment would give a better metabolic control and quality of life.

DETAILED DESCRIPTION:
The current standard of insulin treatment in type 1 diabetes is multiple daily insulin injection therapy (MDII). In the seventies, continuous subcutaneous insulin infusion (CSII) was introduced. CSII has been gaining popularity, perhaps because of technical advances resulting in improved patient comfort. In children five randomised studies(1-5) were completed to compare MDII and CSII. No data were gained about quality of life and impact of disease.

In our trial we focussed on quality of life next to metabolic control.

The trial was an open-labelled,randomised trial. Both efficacy and safety data were collected. The trial started with a 14 weeks run in phase, during all patients started MDII.In the following randomisation phase patients were randomised to continue MDII or to CSII.This phase lasted 14 weeks.In the phase thereafter all patients used CSII for 14 weeks. The trial was concluded by a 14 weeks allocated patient preference phase.

Patients were type 1 diabetic children 4-16 years old with poor metabolic control.hypothesis: better metabolic control in CSII, better quality of life in CSII.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes,
* Diagnosed by the presence of IA-2,
* GAD-65 or islet cell cytoplasmatic auto antibodies,
* Daily insulin adminstration or 1 year of longer,
* Random C-peptide <200 pMol,
* Hba1c>8.0% and/or a history of repeated symptomatic hypoglycaemias,
* Attending regular school

Exclusion Criteria:

* Clinical manifest chronic complications,
* Pregnancy,
* Co-morbidity,
* Mental retardation,
* Psychiatric treatment or symptoms in child or parent,
* Insufficient Dutch language capabilities and absence of telephone at home

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38
Dates: Start 2002-01; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
metabolic control
quality of life

SECONDARY OUTCOMES:
cost effectiveness
surrogate markers for late complications
adverse events
impact of disease

CONTACTS AND LOCATIONS:
Overall Officials: roos Nuboer, MD, Principal Investigator — Erasmus Medical Center; Jan Bruining, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC/Sophia´s children´s Hospital, Rotterdam, Netherlands

REFERENCES:
- [Background] Fox LA, Buckloh LM, Smith SD, Wysocki T, Mauras N. A randomized controlled trial of insulin pump therapy in young children with type 1 diabetes. Diabetes Care. 2005 Jun;28(6):1277-81. doi: 10.2337/diacare.28.6.1277. PMID 15920039
- [Background] Wilson DM, Buckingham BA, Kunselman EL, Sullivan MM, Paguntalan HU, Gitelman SE. A two-center randomized controlled feasibility trial of insulin pump therapy in young children with diabetes. Diabetes Care. 2005 Jan;28(1):15-9. doi: 10.2337/diacare.28.1.15. PMID 15616227
- [Background] Doyle EA, Weinzimer SA, Steffen AT, Ahern JA, Vincent M, Tamborlane WV. A randomized, prospective trial comparing the efficacy of continuous subcutaneous insulin infusion with multiple daily injections using insulin glargine. Diabetes Care. 2004 Jul;27(7):1554-8. doi: 10.2337/diacare.27.7.1554. PMID 15220227
- [Background] Weintrob N, Benzaquen H, Galatzer A, Shalitin S, Lazar L, Fayman G, Lilos P, Dickerman Z, Phillip M. Comparison of continuous subcutaneous insulin infusion and multiple daily injection regimens in children with type 1 diabetes: a randomized open crossover trial. Pediatrics. 2003 Sep;112(3 Pt 1):559-64. doi: 10.1542/peds.112.3.559. PMID 12949284
- [Background] DiMeglio LA, Pottorff TM, Boyd SR, France L, Fineberg N, Eugster EA. A randomized, controlled study of insulin pump therapy in diabetic preschoolers. J Pediatr. 2004 Sep;145(3):380-4. doi: 10.1016/j.jpeds.2004.06.022. PMID 15343195